CLINICAL TRIAL: NCT03727490
Title: The Role of Subscapularis Repair in Reverse Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201611123
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Arthropathy Shoulder
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): This group will have the subscapularis left un-repaired, which is the standard of care for our institution for reverse shoulder arthroplasty.
  Interventions: Other: Standard Treatment
- Study (Experimental): This group will have the subscapularis tendon repaired through a bone to bone repair that will add approximately 5 minutes to the surgical procedure.
  Interventions: Other: Repair

INTERVENTIONS:
Other: Repair — The subscapularis will be repaired.
  Arms: Study
Other: Standard Treatment — No repair will be performed
  Arms: Control

SUMMARY:
The overall goal of the study is to determine if repairing the subscapularis tendon during primary reverse shoulder arthroplasty effects short-term patient outcomes. The study is a patient blinded randomized controlled trial that is currently enrolling.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing primary reverse shoulder arthroplasty

Exclusion Criteria:

* Adults without an intact subscapularis
* Inflammatory arthritis
* Revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons Score | Two Years
  Patient Reported Outcome

SECONDARY OUTCOMES:
Simple Shoulder Test | Two Years
  Patient Reported Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alexander W Aleem, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Department of Orthopaedic Surgery, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No